CLINICAL TRIAL: NCT06941805
Title: Evaluation of Blue and White Collar Employees in Terms of Physical Activity and Physical Fitness (University Example)
Brief Title: Blue and White Collar Employees in Terms of Physical Activity
Status: Completed | Type: Observational
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Other Study IDs: mehmet.sonmez1
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Employees of University; Physical Fitness; Physical Activity
Keywords: Physical Activity; Fitness; Worker; University
MeSH Terms: conditions — Motor Activity | interventions — Physical Fitness; Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- White-collar: Academic and administrative employees of the University
  Interventions: Diagnostic Test: Physical Fitness; Diagnostic Test: Physical activity
- Blue-collar: Technical employees of the University
  Interventions: Diagnostic Test: Physical Fitness; Diagnostic Test: Physical activity

INTERVENTIONS:
Diagnostic Test: Physical Fitness — Physical fitness levels of blue- and white-collar university workers were measured and compared.
Diagnostic Test: Physical activity — Weekly physical activity levels of blue- and white-collar university workers were measured and compared.

SUMMARY:
The aim of our study was to evaluate the weekly physical activity levels and general physical fitness levels of blue-collar and white-collar employees working in a similar field in the university environment.

White-collar employees consisted of academic and administrative staff (n:50) and blue-collar employees consisted of technical service personnel (n:50). In the study, demographic data collection form was used to evaluate demographic data, International Physical Activity Level Questionnaire was used to evaluate physical activity level, 360-degree rotation test was used to evaluate dynamic balance among physical fitness parameters, Short Physical Performance Battery was used to evaluate physical performance, analogue dynamometer was used to evaluate grasp strength, and 30-second sit-to-stand test was used to evaluate muscular endurance.

DETAILED DESCRIPTION:
BACKGROUND: Due to the long hours spent in business life, the nature of the job can affect the physical activity and physical fitness level of individuals. Although some studies have been conducted showing that university employees have low levels of physical activity due to their jobs, there is no study comparing blue- and white-collar university employees whose job descriptions are more similar than in other fields.

OBJECTIVE: The aim of our study was to evaluate the weekly physical activity levels and general physical fitness levels of blue-collar and white-collar employees working in a similar field in the university environment.

METHODS: The present study was of a quantitative nature, with two groups, and was conducted with the participation of academic, administrative, and technical service personnel working throughout the university. The university was located in a developed country with a high income level. A total of 124 university personnel were pre-registered for the study, including 64 academic staff, 60 administrative staff, and 60 technical service personnel. Twenty-four personnel were excluded from the study due to non-compliance with the inclusion and exclusion criteria. The exclusion of ten personnel was due to their advanced age (over 50 years), two due to orthopaedic problems, eight due to non-signing of informed consent, and four due to their occupation as professional athletes. The white-collar employees consist of academic and administrative staff (n: 50), and the blue-collar employees consist of technical service personnel (n: 50).

The study was conducted without the groups meeting each other and without prior knowledge about the measurements. All measurements were performed in a standardized manner and data collected in a single session. The measurements were conducted in suitable areas determined on the university's campus. All measurements were performed by the same researcher to ensure the consistency of the results.

In the study, a demographic data collection form was used to evaluate demographic data, International Physical Activity Level Questionnaire was used for physical activity level, 360-degree rotation test was used to evaluate dynamic balance among physical fitness parameters, and Short Physical Performance Battery (SPPB) was used to evaluate physical performance. Also, the analog dynamometer was used to evaluate grasp strength, and 30-second sit-to-stand test was utilized to assess muscular endurance.

ELIGIBILITY:
Inclusion Criteria:

* being a contracted or permanent staff member of the university
* being between 18-50 years of age, being able to walk independently for 150 meters or more
* having given consent forms to participate in the study voluntarily.

Exclusion Criteria:

* having a health problem that would prevent movement and mobility
* being a professional or amateur licensed athlete
* having taken at least a day off work in the last week.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our sample consisted of blue and white collar personnel working at a university.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Demographic Data | "From October 2023 to June 2024"
  Demographic Data Collection Form was used. This includes such metrics as participant number, age, gender, employment status, working hours, stature, mass, body mass index, smoking habits, and patterns of alcohol consumption.
Weekly Physical Activity Level | "From October 2023 to June 2024"
  The International Physical Activity Questionnaire (IPAQ) is a tool designed to assess levels of physical activity. This scale is a self-report measure of physical activity. The questionnaire in question is designed to assess the level of physical activity undertaken by the subject over the preceding seven days.
Dynamic Balance | "From October 2023 to June 2024"
  The 360-degree rotation test is a methodical procedure that is conducted in accordance with the established protocol. The participant is instructed to step on a marked point with the foot of their choosing. Following a demonstration by the examiner, the participant is instructed to rotate in the direction of their choosing, provided that they do not take a step with their fixed foot. The test is considered complete once the participant returns to the initial position. The duration of the test is recorded by issuing a command to the participant to commence the test. The test is then repeated twice to ensure reliability. Should the total time exceed 3.8 seconds, it is indicated that there is a risk of falling.
Physical performance | "From October 2023 to June 2024"
  The Short Physical Performance Battery (SPPB) is a comprehensive evaluation tool that assesses various aspects of physical performance. The SPPB is composed of three distinct components: firstly, a standing balance test; secondly, a 4-metre walking speed test; and thirdly, a five repetition sit-and-stand test. Each component of the SPPB is assigned a score ranging from 0 to 4, with 0 denoting the inability to perform the test and 4 representing the highest performance category. The maximum attainable score is 12, denoting optimal bodily functionality.
Handgrip strength | "From October 2023 to June 2024"
  Sanlindou 287 Ibs was assessed with a dynamometer from Shanghai, People's Republic of China. The handgrip strength was selected as a preliminary indicator of the global upper extremity muscle strength level. The participants were instructed to grasp the dynamometer in a standard position (sitting position, shoulder adduction, elbow 90 degrees flexed, and forearm in a neutral position) and to attempt to squeeze the device with maximum voluntary contraction. The measurement was repeated three times, and the highest value or average value was recorded.
Lower limb endurance | "From October 2023 to June 2024"
  The 30-second sit-to-stand test is a method of evaluating an individual's lower body strength and endurance. This test is designed to evaluate the participant's endurance in performing sit-ups. The number of sit-ups performed within a 30-second time frame is documented. Participants demonstrating fewer than ten repetitions are considered to have inadequate endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University Health Science Faculty, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was stated in informed consent that the information regarding participant will not be shared to any side.